CLINICAL TRIAL: NCT03176108
Title: Evaluation of a Parent/Child Cognitive-Behaviorial Therapy Program in ADHD Children With Emotional Dysregulation Profile : a Study Prospective, Controlled and Randomized
Brief Title: Evaluation of a Parent/Child Cognitive-Behaviorial Therapy Program in ADHD Children With Emotional Dysregulation Profile
Acronym: DP-KID
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University Hospital, Montpellier (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 9729
Record Dates: First submitted 2017-05-30; First posted 2017-06-05 (Actual); Last update posted 2023-01-23 (Actual); Status verified 2023-01

CONDITIONS: Attention Deficit Disorder With Hyperactivity; Attention-Deficit-Disordered Children
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- CBT Group (Experimental): The CBT group benefits of an intervention based on the program "Better manage its anger and its frustrations" of 15 sessions for the children.
  Parents participate in an CBT intervention of 8 sessions every 15 days. The session allow to develop adapted behaviors, to manage the disruptive behaviors and to improve the relations parents/children.
  Interventions: Behavioral: Cognitive Behavorial Therapy (CBT)
- Control Group (Sham Comparator): The control group participates in an intervention of body mediation (theatre) of 15 session for the children.
  Parents participate in an CBT intervention of 8 sessions every 15 days. The session allow to develop adapted behaviors, to manage the disruptive behaviors and to improve the relations parents/children.
  Interventions: Behavioral: Body mediation

INTERVENTIONS:
Behavioral: Cognitive Behavorial Therapy (CBT) — Cognitive Behaviorial Therapy (CBT)
  Arms: CBT Group
Behavioral: Body mediation — Body mediation (theatre)
  Arms: Control Group

SUMMARY:
Attention Deficit Disorder (ADD) with or without Hyperactivity/Impulsivity (ADHD) is a neurodevelopmental syndrome that has a lasting impact on the child's daily lifestyle and leads to functional impairment. ADHD is recognized as the most common psychiatry disorder in children and it's considered as a public health problem.

ADHD is frequently associated with a new diagnostic entity " Disruptive Disorder with Emotional dysregulation ". This disorder is characterized by crisis of anger with verbal or physical aggression, intensity disproportionate to the context and developmental age.

Few studies have examined the elements of emotional dysregulation in ADHD in children. Many studies have shown the interest of CBT in multimodal management of ADHD symptoms and associated disorders.

The main objective is to evaluate the effectiveness of a Cognitive-Behavioral Therapy Parent/Child program versus a body mediation focused on emotional and behaviorial aspects in ADD children aged 7-13 years with dimensional emotional dysregulation at 6 months after intervention. Secondary objectives are to evaluate the impact of this program, at short-term (at the end of CBT) and at 6 months after intervention, on socio-communicative capacities, quality of life, children's functioning and parental stress.

It's a biomedical research, prospective, controlled, randomized, monocentric, two parallels, with an evaluation of the criteria of blind judgment.

DETAILED DESCRIPTION:
68 patients (parents and children) will be recruited within Montpellier University Hospital. They will be divided into a CBT group and a control group (body mediation).

The CBT group benefits from an intervention based on the program "Better manage its anger and its frustrations" of 15 sessions for the children.

The control group participates in an intervention of body mediation (theatre) of 15 session for the children.

The parents of CBT and Control groups participate in an CBT intervention of 8 sessions every 15 days.

ELIGIBILITY:
Inclusion Criteria:

* Children and adolescents aged 7-13 years ;
* Children with a diagnostic of ADHD (diagnostics criteria from DSM-V);
* Score CBCL-DP ≥ 180 (" Aggressive behavior ", " Anxious-depression " and " Attention problems ") ;
* Children follow-up in Montpellier University Hospital ;
* Parents and children benefit of social security.

Exclusion Criteria:

* Children with a developmental delay or severe language disorder ;
* Families non-french speaking ;
* Absence of consent signed by parents and child ;
* Children not living with at least one parent.

Ages: 7 Years to 13 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 92 (Estimated)
Dates: Start 2017-06-28 (Actual); Primary Completion 2024-03-28 (Estimated); Study Completion 2025-03-28 (Estimated)

PRIMARY OUTCOMES:
Variation between the initial assessment and the month evaluation atfer the end of the intervention on the score of the " Aggressive behavior " subscale at the CBCL (Child Behavior Checklist) | Evaluation at inclusion, 6 months and 12 months
  The Questionnaire is completed by parents

SECONDARY OUTCOMES:
:* Variation of total score on CBCL and score on " Dysregulation profile " (CBCL-DP) on Child Behavior Checklist | Evaluation at inclusion, 6 months and 12 months
  The Questionnaire is completed by parents
Variation of scores on " Strengths and Difficulties Questionnaire " | Evaluation at inclusion, 6 months and 12 months
  Description: The Questionnaire is completed by parents and teachers
Variation of scores on " Parenting Stress Index " | Evaluation at inclusion, 6 months and 12 months
  The Questionnaire is completed by parents
Variation of score on " Beck Depression Inventory " | Evaluation at inclusion, 6 months and 12 months
  The Questionnaire is completed by parents
Variation of scores on " Kidscreen-27 " | Evaluation at inclusion, 6 months and 12 months
  The Questionnaire is completed by parents
Variation of score on " PAR-ENT-Qol " | Evaluation at inclusion, 6 months and 12 months
  The Questionnaire is completed by parents
Variation of score on " Children's Global Assessment Scale " (C-GAS) | Evaluation at inclusion, 6 months and 12 months
  The Questionnaire is completed by the evaluator who receive parents and their child.

CONTACTS AND LOCATIONS:
Overall Officials: Elodie COURTABESSIS, MD PHD, Principal Investigator — University Hospital, Montpellier
Locations (1):
- CHU Montpellier, Montpellier, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Vacher C, Romo L, Dereure M, Soler M, Picot MC, Purper-Ouakil D. Efficacy of cognitive behavioral therapy on aggressive behavior in children with attention deficit hyperactivity disorder and emotion dysregulation: study protocol of a randomized controlled trial. Trials. 2022 Feb 7;23(1):124. doi: 10.1186/s13063-022-05996-5. PMID 35130934